CLINICAL TRIAL: NCT06530758
Title: Does the Format of the Adult ADHD Self-Report Scale Impact the Results: a Randomized Controlled Trial
Brief Title: Does the Format of the Adult ADHD Self-Report Scale Impact the Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: Pro00144202
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASRS without shading and with grouping (Experimental): These participants will receive the ASRS form that does not have shading for the screen positive response options and has the questions grouped (ie, the headings "Part A" and "Part B" will remain on the form).
  Interventions: Other: Altered ASRS format, without shading and with grouping
- ASRS with shading and without grouping (Experimental): These participants will receive the ASRS form that has the screen positive response options shaded and has the questions ungrouped (ie, the headings "Part A" and "Part B" are removed).
  Interventions: Other: Altered ASRS format, with shading and without grouping
- ASRS without shading and without grouping (Experimental): These participants will receive the ASRS form that does not have shading for the screen positive response options and has the questions ungrouped (ie, the headings "Part A" and "Part B" are removed).
  Interventions: Other: Altered ASRS format, without shading and without grouping
- Standard ASRS: with shading and with grouping (No Intervention): These participants will receive the standard ASRS form. This form has the positive response options for each question shaded and has the questions grouped (ie, the headings "Part A" and "Part B" will remain on the form).

INTERVENTIONS:
Other: Altered ASRS format, without shading and with grouping — Participants will be asked to complete the ASRS form without shading and with grouping.
  Arms: ASRS without shading and with grouping
Other: Altered ASRS format, with shading and without grouping — Participants will be asked to complete the ASRS form with shading and without grouping.
  Arms: ASRS with shading and without grouping
Other: Altered ASRS format, without shading and without grouping — Participants will be asked to complete the ASRS form without shading and without grouping.
  Arms: ASRS without shading and without grouping

SUMMARY:
The World Health Organization Adult ADHD Self-Report Scale v1.1 (ASRS) is frequently used in family medicine clinics to screen for ADHD. Numerous studies have found the ASRS has a low positive predictive value. Compounding this concern is the format of the ASRS. Specifically, the answers on the ASRS that lead to screen positive results are shaded in gray and grouped together, which may make it easy for patients to discern which responses should be selected for a positive screen.

DETAILED DESCRIPTION:
The ASRS is used widely to screen for ADHD in adults. It has 18 questions, with response options "never," "rarely," "sometimes," "often," and "very often." The 6 questions considered most predictive of ADHD are grouped together in Part A and questions that are meant to provide additional cues are grouped together in Part B. The options that are considered a positive response vary between questions; for some questions the option is at least "sometimes," while for others it is at least "often." The positive response options are shaded on the ASRS. A person is considered to have a positive screen if 4 of the 6 questions in Part A are positive.

The objective of this trial is to determine if the shading and grouping on the ASRS impacts screening results. This trial has a 2x2 factorial design set in a family medicine clinic(s). When a patients check in for an appointment, clinic staff will offer them a survey that includes 1) demographic questions and 2) 1 of the 4 versions of the ASRS, the version they receive is randomized (with programming). Most patients will take approximately 5 minutes to complete the survey prior to them seeing the family physician.

ELIGIBILITY:
Inclusion Criteria:

* 19 - 65 years old
* Patients who are registering for their appointment at the family medicine clinic
* Patients who are expected to be in the reception area for ≥5 minutes before going to a clinic room

Exclusion Criteria:

* Any patients who do not have the capacity to complete the form (e.g., cognitive impairment, unable to read English, unable to use a computer)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Screen positive rate | Through study completion, estimated to be 2 months
  Poisson regression to determine the relative risk of a screen positive among the different versions of the form. We will include the following covariates: shading, grouping, shading x grouping, suspect ADHD without diagnosis, ADHD diagnosis, sex, and age.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Kraut, Principal Investigator — University of Alberta
Locations (1):
- Shifa Medical Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraut RY, Ono C, Garrison S, Kamal O, Doroshuk ML, Vandermeer B, Amanna G, Babenko O. Does the format of the adult ADHD self-report scale influence screen-positive rates? A randomized controlled trial in primary care. Front Psychiatry. 2026 Jan 2;16:1646293. doi: 10.3389/fpsyt.2025.1646293. eCollection 2025. PMID 41551194